CLINICAL TRIAL: NCT00216281
Title: Correlation of Phenotype, Genotype and Clinical Efficacy/Toxicity of Clozapine Augmented by Atomoxetine for Treatment Refractory Schizophrenia (CAPG Study)
Brief Title: Efficacy and Safety Study of Clozapine Augmented by Atomoxetine Versus Clozapine Augmented by Placebo in Patients With Chronic Resistant Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Hoffmann-La Roche (Industry); Shekhar, Anantha M.D., Ph.D. (Individual)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0501-47
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Clozapine; Atomoxetine
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- clozapine with AZT added (Active Comparator): Clozapine augmented with Atomoxitine up to 40mg
  Interventions: Drug: Clozapine augmented with atomoxetine up to 40 mg or placebo
- placebo (Placebo Comparator): Subjects will have a placebo pill added to their clozapine regimen.
  Interventions: Drug: Clozapine augmented with atomoxetine up to 40 mg or placebo

INTERVENTIONS:
Drug: Clozapine augmented with atomoxetine up to 40 mg or placebo

SUMMARY:
This is a randomized, placebo-controlled study to assess the efficacy and safety of ATX augmentation of CLZ as a treatment for the cognitive symptoms of schizophrenia. A total sample size of 126 subjects diagnosed with schizophrenia and being treated with the antipsychotic clozapine will undergo genotyping. These subjects will have an initial assessment at four weeks and regular follow-up assessments for a total period of 52 weeks. These subjects will be randomized to continued treatment with CLZ and augmentation with ATX or Placebo.

DETAILED DESCRIPTION:
The purpose of this study is to scientifically explore the potential of pharmacogenetic applications as a means of predicting the clinical efficacy and safety of treatment with clozapine and atomoxetine in a treatment resistant schizophrenic population.

The principle enzyme involved in the metabolism of clozapine is CYP1A2 with minor contributions from CYP2D6. However, all the subjects will be on a stable dose of clozapine and will continue on the same dosage throughout the study. On the other hand, half the number of subjects will be randomized to augmentation with atomoxetine and since atomoxetine is predominantly metabolized by CYP2D6 with contributions from CYP2C19, we will focus on genetic variations for CYP2D6 and CYP2C19.

The goal of this study is to associate atomoxetine and metabolite drug concentrations with clinical efficacy and the development of any clinical adverse drug reactions and to determine whether clinical outcome (efficacy and ADRs) experienced following drug ingestion are more likely to be seen in patients who manifest CYP2D6 and/or CYP2C19 polymorphism(s). Other indications for pharmacogenetics in patient care, relevance of therapeutic drug monitoring, augmentation strategies and dosage guidelines may be generated from the experience and results of this study.

Primary Objectives

1. To compare the effects of the combination of CLZ+ATX on cognitive function in patients with schizophrenia, as measured by change in a Composite Cognitive index derived from a battery composed of standardized cognitive tests, the Brief Assessment of Cognition in Schizophrenia..
2. A total sample of 126 subjects diagnosed with schizophrenia and being treated with the antipsychotic clozapine, will be recruited to participate in the study. All 126 subjects will undergo genetic testing after obtaining informed consent, for 31 known mutations in CYP2D6 including gene duplication and deletion as well as, two mutations in CYP2C19.

Secondary Objectives

1. Determine the concentration of atomoxetine and its two prominent metabolites (4-hydroxyatomoxetine, and N-desmethylatomoxetine) at the end of week one and four weeks after initiating therapy by LC/MS/MS analysis.
2. Obtain weekly complete blood counts and CLZ levels on screening, at the end of week one and week four.
3. Clinically evaluate patients and document any adverse drug reactions that occur after starting treatment with atomoxetine
4. To examine the effects of the combination of CLZ+ATX on psychopathology as measured by the Positive and Negative Syndrome Scale (PANSS) scores (PANSS Total, PANSS Positive, PANSS Negative), the Montgomery-Asberg Depression Rating Scale and the Clinical Global Impressions-Improvement Scale
5. To examine the effects of the combination of CLZ+ATX on measures of social cognition: Penn Emotional Recognition and Facial Memory Tests.
6. To compare the effects of the combination of CLZ+ATX on weight change from baseline.
7. To examine the effects of the combination of CLZ+ATX on daily functioning as measured by the NOSIE.
8. To examine the effects of the combination of CLZ+ATX on extrapyramidal signs and motor symptoms as measured by the Barnes Akathesia Rating Scale (BARS), the Abnormal Involuntary Movement Scale (AIMS), and the Simpson-Angus Scale (SAS).
9. To evaluate the safety of the combination of CLZ+ATX as measured by treatment-emergent adverse events and changes in vital signs, clinical laboratory analytes, and electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Schizophrenia that meets the diagnostic criteria as defined in the Diagnostic and Statistical Manual of Mental Disorders (4th edition, text revision) (DSM-IV-TR), APA 2000).
2. Adult (18-65) males or females with a confirmed primary diagnosis of schizophrenia.
3. Stable symptoms as determined by a score of 70 or less on the PANSS.
4. Women of child bearing potential must be using a medically accepted means of contraception.
5. Adequate cognitive function (IQ > 65) as assessed by the WRAT3, with a level of understanding sufficient to perform all tests and examinations required by the protocol.
6. Considered reliable.
7. Stable on clozapine treatment. Criteria for stability defined as follows:

   * Patients should have been taking oral clozapine daily for the last 4 weeks (with no change in clozapine dose in the 4 weeks prior to screening).
   * Patients must not require chronic add-ons or have taken "as needed" antipsychotic or antidepressant medications in the last four weeks to control agitation, behavioral disturbance, or primary psychiatric symptomatology.
   * There must have been no significant change in the level of care required, caused by worsening of schizophrenia in the last four weeks. For example any escalation from lesser to greater intensity of treatment or ER visits.
   * Patients must not be taking any additional psychotropic medications including health food supplements judged by the investigator to be likely to have central nervous system activity (for example, St. John's Wort, ginkgo biloba leaf, melatonin).
   * Patients must not have received a depot antipsychotic within the past 8 weeks days.
8. Each patient must be judged competent and able to understand the nature of the study and must sign an informed consent document prior to participation in the study.
9. Patients must be able to swallow medications.

Exclusion Criteria:

1. Clinically significant organic disease that, in the opinion of the investigator, would put the patient at significant risk from study procedures or interfere with data interpretability. This includes hepatic (specifically any degree of jaundice), renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, or immunologic conditions.
2. Potentially serious or unstable medical condition that is likely to require excluded medications or other significant treatment during the course of this treatment.
3. Patients who have not tolerated atomoxetine in the past or have history of clinically significant adverse effect(s) during prior treatment with atomoxetine.
4. Patients who have not tolerated oral CLZ in the past or experienced significant adverse effect(s) in the past.
5. History of non-response to clozapine (treatment refractory) defined as unambiguous lack of improvement despite contiguous adequate trial of at least 14 weeks of treatment.
6. Clozapine blood levels outside the optimum CLZ plasma levels of 350 to 400 ng/ml.
7. Women who are pregnant, breastfeeding, or refuse to use adequate birth control.
8. Significant risk of suicidal behavior or pose an imminent significant threat to others, at the time of screening.
9. History of alcohol or drug dependence (except nicotine and caffeine) that meets DSM IV criteria, within the past six months or have a history of drug or alcohol abuse within the past 30 days. Patients who have history of cannabis use for recreational purposes may be enrolled if in the opinion of the PI, the drug use pattern is not primarily related to a psychiatric condition or diagnosis.
10. Have abnormal blood pressure in the opinion of the investigator.
11. Electrocardiograms (ECGs) outside the normal limits.
12. Abnormal clinical laboratory test results outside the normal range.
13. History of agranulocytosis (absolute neutrophil count <500 mm3).
14. Uncorrected hypothyroidism, hyperthyroidism or abnormal thyroid-stimulating hormone (TSH) concentrations. Patients previously diagnosed with hyperthyroidism or hypothyroidism who have been treated on a stable dose of thyroid supplement for at least 3 months, have medically appropriate TSH concentrations, and who are clinically euthyroid are allowed.
15. History of clinically significant head injury.
16. History of allergic reaction to clozapine or atomoxetine or any condition that could be aggravated by treatment with these medications (for example, narrow-angle glaucoma, urinary retention or hesitancy).
17. one or more seizures without a clear and resolved etiology.
18. Hearing or visual impairment severe enough to interfere with performance on cognitive tests.
19. Patients who have taken a monoamine oxidase inhibitor (MAOI) drug (for example Nardil™, Parnate™, or Eutron™ for depression) or tryptophan within the last 2 weeks prior to screening.
20. History of electroconvulsive therapy within the previous year.
21. History of mental retardation.
22. Have grade-level equivalent score of less than 8th grade as determined by WRAT3. This means that a patient must have a raw score of 40 or above (IQ equivalent of 81) in order to qualify.
23. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
24. Investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
25. Patients who, in the opinion of the investigator, are unsuitable in any way to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Impact of treatment will be based on clinical examination, laboratory values, and rating scales including, PANSS, CGI, AIMS, BAS, SAS, cognitive measures, NOSIE. | 375 days
  Via rating scales and cognitive measures, effects of CLZ and ATZ on congitive function will be assessed. A total of 126 suybjets diagnosed with Schizophrenia will be recruited, consented, and treated with CLZ and ATZ. They will undergo genetic testing for 31 mutations of CYP2D6 including gene duplication and deletion as well as, two mutations in CYP2C19.

SECONDARY OUTCOMES:
Concentrations | week 1 and week 4
  Determine the concentration of atomozetine and its two prominent metabolites
blood cell counts | week 1 and week 4
  Obtain complete blood counts and CLZ levels on screening and at week 1 and 4
adverse events | day one forward
  clincal evaluation for adverse drug interactions that occur with the start of atomoxetine
symptom measure | screen, day 1 and all f/u visits
  Panss, MADRS and CGI scales completed at each visit
social cognition | screening, day 1 and f/u visits
  assessment of cognitive function via Penn Emotional REcognition and facial memory tests.
weight change | day one and follow up visits
  measures of weight change from baseline.
daily functioning | baseline through f/u visits
  measure of daily functioning via the NOSIE and extrapyraminal/motor signs via the BARS and AIMS scales
adverse events 2 | baseline forward
  evaluation via vital signs, clinical labs and ECG for safety

CONTACTS AND LOCATIONS:
Overall Officials: Anantha Shekhar, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- LaRue Carter Hospital, Indianapolis, Indiana, United States